CLINICAL TRIAL: NCT02016378
Title: EEG/Event-related Brain Potential Risk Markers as Predictors and Outcomes of SUD Treatment in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Maryland (Other)
Responsible Party: Principal Investigator, Brian Hicks, Research Assistant Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 655655; R03DA034718 (NIH)
Record Dates: First submitted 2013-11-21; First posted 2013-12-20 (Estimated); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham retraining (Sham Comparator): Participants in this condition will participate in a computerized task wherein the size of pictures of drug and non-drug related stimuli are increased or decreased based on the tilt (left or right) of the pictures, but without regard to the content (i.e., drug or non-drug).
  Interventions: Behavioral: Sham retraining
- Bias retraining (Active Comparator): Participants in this condition will participate in 6 sessions of a computerized bias retraining.
  Interventions: Behavioral: Bias retraining

INTERVENTIONS:
Behavioral: Bias retraining — Participants will view pictures of drug (e.g., alcohol) and non-drug stimuli (e.g., soft drinks) on a computer. Participants will then use the computer to make the drug pictures smaller and the non-drug pictures larger.
  Arms: Bias retraining
Behavioral: Sham retraining — Participants will view pictures of drug and non-drug related stimuli on a computer. Participants will then use the computer to make the pictures larger or smaller based on the tilt of the picture (slightly to the left or right), but without regard to the content of the picture.
  Arms: sham retraining

SUMMARY:
This study investigates the effect of a computerized approach/avoidance retraining (aka cognitive bias modification) over and above treatment as usual for patients in treatment for substance use disorders. The computerized training entails viewing pictures of drug and non-drug related stimuli, and then using the computer to make the drug pictures smaller and the non-drug pictures larger. Participants will also take part in an EEG/event-related brain potential assessment at the beginning and end of treatment to identify brain measures that are associated with treatment response.

DETAILED DESCRIPTION:
Methodology Participants must be receiving treatment for substance use disorders in the adolescent program of the University of Michigan Addiction Treatment Services (UMATS) clinic. Participants must be between the ages of 14-65.

The study entails five components

1. Neurophysiological assessment. (Baseline)
2. Assessment of substance use and psychiatric disorders. (Baseline)
3. Bias retraining treatment protocol. (after baseline, 6 training sessions over a two week period)
4. Second neurophysiological assessment at the end of treatment. (6 weeks after baseline)
5. Six-month follow-up to assess substance use and psychiatric disorders. (6 months after baseline)

Each component is described in more detail below:

1. Assessment of substance use and psychiatric disorders will be completed using well-validated structured interviews and questionnaires. This assessment will take place as soon as participants can be scheduled following their entry into treatment at the UMATS clinic.
2. Neurophysiological assessment will entail several procedures that reliably elicit brain responses that are associated with substance use disorders and antisocial behavior. The first neurophysiological assessment will take place as soon as participants can be scheduled following their entry into treatment at the UMATS clinic.

The different tasks are described below. Participants will be asked to perform tasks that involve responding to letters and pictures on a computer monitor while physiological responses will be recorded continuously during the experiment. This will be achieved by the use of sensors positioned on the head, forearms, palms, and face. These sensors are filled with a nonirritating paste and attached to the skin using medical tape.

The tasks are as follows:

1. Picture Viewing and Emotion Regulation Task-Duration: approximately 40 minutes The subject will be presented with a number of different pictures from the International Affective Picture System (IAPS) including traditional unpleasant, neutral, and pleasant images as well as images of drugs and drug-related paraphernalia. Pictures are presented following an instruction cue asking the person to enhance (upregulate) or diminish (downregulate) their affective responses.
2. Go/No go task - Duration: 10 minutes During this procedure, participants will respond to two different letters by selecting one of two buttons that are associated with each letter. They will be asked to inhibit their response if the letter they are viewing is the same as the letter just viewed. It is intended to measure cognitive control. Drug-related pictures will also be included as distractors to examine their effects on performance and EEG/event-related potential (ERP) measures.
3. Gambling/feedback task-Duration: 10 minutes During this procedure, participants will see 2 squares, side-by-side on the monitor in front of them. Each square will have a money amount displayed inside of it. Sometimes the squares show 5 cents, and sometimes they show 25 cents. The task is simply to choose one of the squares on each trial, either the one on the left or the one on the right. After a delay of about one second, the participant will be told if he or she won or lost the amount of money inside the square he or she chose. If the selected square turns GREEN that means the participant won the amount of money shown inside the square. If the chosen square turns RED that means the participant lost the amount of money shown inside the square. At the same time, the unselected will also turn either green or red, to inform the participant how much he or she would have won or lost if the other square had been selected.

3) Bias retraining treatment protocol. In addition to treatment as usual at the UMATS clinic, participants will be randomized into either bias retraining or sham training conditions. At a pre-test session, participants will complete an approach-avoidance task (AAT) to measure initial bias to drug-related stimuli. The AAT are each completed on a laptop computer.

The AAT includes 20 pictures of drug-related stimuli and 20 pictures of non-drug related stimuli. Pictures are presented equally in landscape and portrait format. After the pictures appear on a monitor, participants will be instructed to use a joystick to either enlarge (pull the joystick closer) or shrink (push the joystick away) the pictures. In this task, the required response is unrelated to the content of the pictures. Specifically, participants are instructed to pull the joystick to approach pictures in portrait format or push pictures in landscape format. The difference between the median response time for drug versus non-drug related pictures is used as a measure of bias. The AAT takes 5 minutes to complete.

The bias retraining protocol will then utilize the AAT. Participants will again be instructed to push or pull the joystick dependent upon whether the picture is in portrait or landscape formant. For participants in the experimental condition, all drug-related pictures will be in landscape format, that is, all participants in the experimental condition will push the joystick to shrink the drug-related pictures. For participants in the control condition, drug-related pictures will be presented equally in portrait and landscape format. During training, participants have to correct all errors. Training sessions will entail 200 trials with a short break at the halfway point. Each session takes about 15 minutes to complete.

The pre-test assessment of bias (AAT) will take place as soon as participants can be scheduled following their entry into treatment at the UMATS clinic. The bias retraining protocol will begin the day following the pre-test assessment of bias. Participants will then take part in 6 training sessions (each requires approximately 15 minutes to complete) over a two week period.

Prior to and following each administration of the AAT, participants will complete a rating of their current feelings of craving to use drugs on a 6-point scale ranging from I don't want to use drugs at all to I would love to use drugs right now. If the participant endorses a 4 or higher on the scale following presentation of the AAT, they will be queried by research staff who will be trained in basic cognitive behavioral techniques to assist the participant in reducing any feelings of craving. As participants are actively engaged in treatment for substance use problems (i.e., consistently thinking and talking about drug use), it is unlikely that words or pictures of drug-related stimuli will elicit sufficient craving to trigger a relapse. Also, all participants will either be in the presence of or near a parent and/or regular treatment provider, further minimizing the risk that any procedures would elicit a relapse.

Participants will also complete a brief symptom inventory at their bias retraining sessions so that we can track their progress over the course of treatment. The participant's primary therapist will also be asked to make brief ratings regarding the participant's engagement and progress at the end of active treatment. Finally, to provide an objective measure of treatment adherence, participants will be drug tested. Drug testing is conducted randomly as part of UMATS treatment, and we will request access to the results of those tests.

4) A second neurophysiological assessment will take place 6 weeks following the baseline assessment, at which point participants will have transitioned out of active treatment (e.g., intensive outpatient). Participants will repeat the same protocol as the first neurophysiological assessment in order to detect any changes in brain responses as a consequence of treatment condition. Participants will also complete the AAT and a brief inventory of symptoms.

5) Six months after entry into treatment at UMATS, participants will be asked to complete questionnaires regarding their substance use and psychiatric symptoms as well as the AAT.

Statistical Design We predict that symptom measures and EEG/ERP measures assessed at baseline will be associated with treatment response as measured by scores on the brief symptom inventory administered at training sessions, results of drug testing, and therapist ratings. Multilevel models will be used to estimate the associations between baseline measures (modeled as fixed effects) and the repeated measures of the outcome variables (repeated measures nested within individuals). To examine the effects of treatment condition (bias retraining versus sham training), a group-based multilevel model (similar to repeated measures ANOVA) will be used to test for any group differences on the EEG/ERP measures assessed at baseline and the follow-up neurophysiological assessment. Similar group-based multilevel models (similar to repeated measures ANOVA) will also be used to test for group differences on the substance use and psychiatric symptom measures assessed at baseline and the 6-month follow-up, as well as the measures of treatment progress (drug tests, symptom measures, therapist ratings) assessed between the baseline assessment and the second neurophysiological assessment at the end of treatment.

Power analysis and target N for recruitment. For the regression and multilevel modeling analysis of dimensional outcomes, an n = 85 will provide 80% to detect the anticipated effect (r = .30, α = .05). For the group-based multilevel models, groups of 41 will provide 80% to detect the anticipated effect. Therefore, our goal is to recruit enough participants such that each group (experimental and control) will include at least 40 participants with a baseline and follow-up neurophysiological assessment. We anticipate a 15% attrition rate. Therefore, we plan to recruit 94 participants.

ELIGIBILITY:
Inclusion Criteria:

Patient in treatment for substance use disorders. Alcohol use problems. -

Exclusion Criteria:

Detoxification treatment. Severe mental illness (e.g., psychotic symptoms)

-

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in Youth Outcome Questionnaire-Self-report scores | baseline, 6 weeks and 6 months after the start of treatment
  This instrument is used to track symptoms throughout treatment. It will be used at baseline, 2x week for 2 weeks, 6 weeks from baseline (end of treatment), and at a 6 month follow-up assessment. The primary outcome is the growth curve of the scores over time.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hicks, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Addiction Research Center, Ann Arbor, Michigan, United States